CLINICAL TRIAL: NCT07324148
Title: Acupuncture for Erectile Dysfunction Among Patients With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: a Clinical Trial
Brief Title: Acupuncture for Erectile Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Attending doctor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025_267_KY
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS); Erectile Dysfunctions; Acupuncture
MeSH Terms: conditions — Erectile Dysfunction | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental)
  Interventions: Device: Acupuncture
- Sham acupuncture group (Sham Comparator)
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — Sanyinjiao (SP6), Zhongliao(BL33), Shenshu(BL23), Huiyang(BL35), Guilai(ST29), Guanyuan(CV4), Shenmen(HT7) and Baihui(GV20) are selected as acupoints protocol. Acupuncture treatment consists of 20 sessions over an 8-week period (3 sessions in each of the first 4 weeks, and 2 sessions in each of the remaining 4 weeks).
  Arms: Acupuncture group
Device: Sham acupuncture — The participants in the sham acupuncture group will receive sham acupuncture treatment in SP6, BL33, BL23, BL35, ST29, HT7, CV4, and GV20. The duration and frequency of sessions are the same as in the acupuncture group.
  Blunt needles will be inserted through the fixed pad to reach the surface of the skin without piercing. Needles will be lifted, thrusted and twirled gently for 3 times to simulate the effects of the needle tip penetrating the skin.
  Arms: Sham acupuncture group

SUMMARY:
Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS) is a prevalent chronic urological disease. CP/CPPS severely impacts patients' quality of life. It is characterized by recurrent pelvic floor pain, lower urinary tract symptoms, and often accompanied by psychological issues and sexual dysfunction (duration ≥3 months, no confirmed infection/pathology).

The investigators have completed a large-sample, multi-center randomized controlled trial (RCT) involving 440 patients with CP/CPPS before. The clinical trial confirmed the sustained efficacy of acupuncture for the symptoms of pain, lower urinary tract symptoms, and anxiety and depression among patients with CP/CPPS. However, the trial revealed no significant improvements in sexual dysfunction in the acupuncture group compared to the sham acupuncture group after 8 weeks of treatment.To address this limitation, the current study is designed, which aims to optimize the clinical acupuncture protocol for CP/CPPS and evaluate whether it can enhance outcomes for psychogenic erectile dysfunction (ED) associated. Additionally, mass cytometry and liquid suspension chip technology will be used to explore systemic and local immune mechanisms underlying acupuncture's effects for CP/CPPS. Functional magnetic resonance imaging (fMRI) and metabolomics will be integrated to analyze patients' systemic states from central nervous system and metabolic perspectives, comprehensively elucidating the multi-dimensional mechanisms by which acupuncture alleviates CP/CPPS.

ELIGIBILITY:
Inclusion Criteria:

* Conforms to the diagnosis of CP/CPPS and pED at the same time;
* Aged between 18-50 years old;
* 8≤IIEF-5 score≤21
* Have a fixed sexual partner and a regular sexual intercourse of ≥1 time/week during treatment period;
* Voluntarily sign an informed consent form.

Exclusion Criteria:

* Patients with drug-induced or organic ED.
* The existence of lesions that may affect erectile function, such as penile cancer, penile sclerosis, penile anatomical deformity, testicular cancer, urinary system stones or neuropathy, etc.
* History of trauma or surgery in pelvic region.
* Patients with hypogonadism.
* Usage of drugs or therapies that relieve CP/CPPS or ED symptoms in the previous 1 month.
* Have received hormonal or psychiatric drugs in the previous 3 months.
* Bladder outlet obstruction, overactive bladder, neurogenic bladder, interstitial cystitis, glandular cystitis, sexually transmitted diseases, bladder tumors, prostate cancer, penile cancer, penile stone, other types of prostatitis.
* With a residual urine ≥100ml.
* Symptomatic urinary tract infection.
* Diseases affecting the function of the lower urethra, such as multiple sclerosis, senile dementia, Parkinson's disease, spinal cord injury, caua equina nerve injury, stroke and multisystem atrophy, etc.
* Severe diseases in heart, lung, brain, liver, kidney and hematopoietic system , mental illness and obvious cognitive function disorders.
* Patients with poor compliance

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the International Erectile Function Index-5 (IIEF-5) score | Week 8
  IIEF-5 is a short verified scale used to evaluate erectile function. It Includes 5 items, with each item ranging from 1-5 points. The total score of IIEF-5 ranges from 5-25 points, with 21-25 indicating normal, 12-21 mild disorder, 8-11 moderate disorder and 5-7 severe disorder.

SECONDARY OUTCOMES:
The change from baseline in the International Erectile Function Index-5 (IIEF-5) score | Weeks 4, 20 and 32.
  IIEF-5 is a short verified scale used to evaluate erectile function. It Includes 5 items, with each item ranging from 1-5 points. The total score of IIEF-5 ranges from 5-25 points, with 21-25 indicating normal, 12-21 mild disorder, 8-11 moderate disorder and 5-7 severe disorder.
Change from baseline in the Erection Hardness Score (EHS). | Weeks 4, 8, 20 and 32
  The verified single-entry EHS scale is used to evaluate the hardness of the penis in sexual life. It ranges from 0 to 4. 0 refers to penis does not enlarge; 1 refers to penis is larger, but not hard 2 Penis is hard, but not hard enough for penetration 3 Penis is hard enough for penetration, but not completely hard 4 Penis is completely hard and fully rigid
Proportion of patients with a reduction of ≥6 points from baseline in the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) total score. | Weeks 4, 8, 20 and 32
  NIH-CPSI consists of 13 items, which are organized into three domains of pain, urinary symptoms, and quality of life impact. The total score of NIH-CPSI ranges from 0 to 43, with higher scores indicating more severe symptoms.
Change from baseline in the International Prostate Symptom Score (IPSS) score. | Weeks 4, 8, 20 and 32
  The IPSS assess the severity of lower urinary tract symptoms in men. The total score of IPSS ranges from 0 to 35, with higher scores indicating more severe symptoms.
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) score. | Weeks 4, 8, 20 and 32
  The HADS is a 14-item scale to screen for anxiety and depression. The total score of HADS ranges from 0 to 42, with higher scores indicating more severe anxiety and depression
Change from baseline in the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) and VAS scores. | Weeks 4, 8, 20 and 32
  The EQ-5D-5L is used to measure health-related quality of life. It consists of a descriptive system and a visual analogue scale (VAS). The descriptive system includes dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A health state utility score can be derived using population-based value sets. The VAS component asks patients to rate their overall health on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Assessment of patient expectations for acupuncture. | Baseline
  Patients will be asked that what do you expect your erectile dysfunction will be in 8 weeks.
The proportion of participants rates their overall improvement as "very much improved" or "much improved" based on the Patient Global Impression-Change (PGI-C) | Weeks 8 and 32
  The Patient Global Impression-Change (PGI-C) is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse" or "very much worse".
Patient Assessment of Blinding Effectiveness | Within 5 minutes after any acupuncture session in Week 8.
  Patients are asked whether they have received traditional acupuncture.

OTHER OUTCOMES:
Safety assessment | Weeks 1-32
  The adverse events will be recorded throughout the trial, whether related to the treatment or not.
Combination treatment | Weeks 1-32
  Combination treatment used throughout the trial will be documented
Changes in peripheral immune cell types | Baseline, Week 8.
  Employed proteomics-based mass cytometry technology are used to obtain the overview of the changes in peripheral immune cell types in venous blood and prostatic fluid.
Change in the immune phenotype spectrum of CP/CPPS patients | Baseline, week 8
  Liquid suspension chip technology will be used to detect the levels of cytokines in serum and prostatic fluid, and establish an organic connection between the changes in prostatic fluid cytokine protein levels and the expression changes of tissue immune-related genes.
Central mechanism underlying the effects of acupuncture for CP/CPPS and ED | Baseline, week 8
  Functional magnetic resonance imaging will be used to analyze the effects of acupuncture to reveal the central mechanism
Urine metabolism | Baseline, week 8
  Metabolomics (urine) will be analysed to provide a more profound analysis at the metabolic level to reveal the mechanism of acupuncture.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until until six months after publication.
Access Criteria: Formal request should be sent to the author (puzhisun@163.com) with a methodologically sound proposal. Researchers whose proposal has been approved will sign a data access agreement